Statistical Analysis Plan – OS Follow-up addendum

Study Code D699BC00001

Edition Number 2.0

Date 3 May 2022

A Randomised, Double-blind, Parallel-group, Multicentre, Phase III Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX<sup>TM</sup>) 500 mg with Anastrozole (ARIMIDEX<sup>TM</sup>) 1 mg as Hormonal Treatment for Postmenopausal Women with Hormone Receptor-Positive Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Been Treated With Any Hormonal Therapy (FALCON)

A Randomised, Double-blind, Parallel-group, Multicentre, Phase III Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX<sup>TM</sup>) 500 mg with Anastrozole (ARIMIDEX<sup>TM</sup>) 1 mg as Hormonal Treatment for Postmenopausal Women with Hormone Receptor-Positive Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Been Treated With Any Hormonal Therapy (FALCON)

| Global Product Statistician | | |
|-----------------------------|-----|------|
| | PPD | Date |

| Signature o | f Global Product Statistician | 2 |
|-------------|---------------------------------------------------------|----|
| TABLE OF | CONTENTS | 3 |
| List Of Abl | previations | 4 |
| amendment | history | 5 |
| 1. Study | Details | 6 |
| 1.1 St | udy objectives | 6 |
| 1.2 St | udy design | 6 |
| 1.3 No | umber of subjects | 6 |
| 2. Analy | sis Sets | 6 |
| 2.1 V | olations and deviations | 6 |
| 3. Follov | v-up outcome variables | 7 |
| 3.1 D | isposition and anti-cancer therapy variables | 7 |
| 3.2 O | verall survival | 7 |
| 3.3 Be | est response to first subsequent breast cancer therapy | 7 |
| 3.4 Sa | ıfety | 7 |
| 3.5 Ex | aposure to study drug | 7 |
| 3.6 Q | uality of Life (QoL) questionnaires | 7 |
| 4. Analy | sis Methods | 7 |
| 4.1 G | eneral principles | 7 |
| 4.1.1 | Multiple testing strategy | 8 |
| 4.2 A | nalysis methods | 9 |
| 4.2.1 | Disposition and anti-cancer therapy | 9 |
| 4.2.2 | Overall survival | 10 |
| 4.2.3 | Best response to first subsequent breast cancer therapy | 12 |
| 4.2.4 | Exposure to study drug | 14 |
| 4.2.5 | Safety | 14 |
| 4.2.6 | Quality of Life (QoL) questionnaires | |
| 5 Refere | ences | 17 |

# LIST OF ABBREVIATIONS

| Abbreviation or special term | Explanation |
|---|---|
| DCO | Data cut off |
| FACT-B | Functional Assessment of Cancer Therapy – Breast |
| ITT | Intention to Treat |
| ORR | Objective response rate |
| OS | Overall Survival |
| PFS | Progression-free survival |
| PT | Preferred term |
| QoL | Quality of Life |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SOC | System organ class |
| TLFs | Tables, listings, and figures |
| TOI | Trial Outcome Index |

# AMENDMENT HISTORY

| Date | Brief description of change |
|---|---|
| 20 October 2017 | First draft – addendum to SAP Edition 3 (27 April 2016) |
| 3 May 2022 | Second draft – per protocol version 6.0 (17 December 2021), change of final overall survival (OS) analysis trigger from when 75% of patients have died to: when at least 65% of patients have died and at least 8 years have passed since the last patient was enrolled; summaries of data on protocol deviations and concomitant medication are also generated; retain OS TLF original numbering and add a suffix for OS analysis |

### 1. STUDY DETAILS

# 1.1 Study objectives

The only objective of the study relevant to the overall survival (OS) follow-up analysis is the secondary objective:

To compare the OS of patients treated with fulvestrant 500 mg versus patients treated with anastrozole 1 mg.

## 1.2 Study design

The study design relevant to the OS is as follows:

After the data cut-off for the primary progression-free survival (PFS) analysis, all the remaining patients, regardless of whether they are still receiving randomised treatment, will enter the survival follow-up phase. An interim analysis of OS data will be performed at the time of the PFS analysis and an updated survival analysis will be performed when at least 65% of patients have died and at least 8 years have passed since the last patient was enrolled, July 11, 2014. After the updated survival analysis, data collection will cease for this study and the patient's treatment will be unblinded.

## 1.3 Number of subjects

The sample size calculations are described in the main SAP.

### 2. ANALYSIS SETS

All patients, defined as everyone who signed informed consent, will be used to summarise patient disposition.

The Intention to Treat (ITT) analysis set, as defined in the main SAP, will be used to analyse OS, and to summarise post-discontinuation anti-cancer therapy, important protocol deviations, concomitant medications, best overall tumour response to first subsequent therapy, Quality of Life (QoL) questionnaires: Functional Assessment of Cancer Therapy – Breast (FACT-B) and EQ-5D.

The Safety analysis set as defined in the main statistical analysis plan (SAP), will be used to summarise serious adverse events (SAE), deaths and exposure.

#### 2.1 Violations and deviations

Important protocol deviations post the data cut-off (DCO) for the primary PFS analysis will be summarised and listed by treatment group.

#### 3. FOLLOW-UP OUTCOME VARIABLES

# 3.1 Disposition and anti-cancer therapy variables

Patient disposition is defined as the number of patients who enrolled; randomised; received treatment, or not; continued to receive treatment, or not, at DCO for the updated OS analysis; were ongoing, or terminated, at DCO.

Post-discontinuation disease-related anticancer therapy is defined as the medications recorded on the Post-Withdrawal Cancer Therapy (CAPRXPOST) CRF page.

Concomitant medications will be listed and summarised by treatment group for the survival follow-up phase.

#### 3.2 Overall survival

Overall survival is defined in section 3.2.1 of the main SAP.

## 3.3 Best response to first subsequent breast cancer therapy

Best response to first subsequent cancer therapy, as collected on the Post-Withdrawal Cancer Therapy CRF page, will be summarised overall and by type of therapy.

## 3.4 Safety

Deaths and SAEs are the only safety variables to be summarised in the Follow-up analysis, as described in section 3.3 of the main SAP.

# 3.5 Exposure to study drug

Derivations of exposure to study drug remain unchanged from the PFS analysis, specifically total duration of fulvestrant will be derived, in months, as follows:

{[earliest of (last dose date +28) or death date] – first dose date +1} / (365.25/12)

Total duration of anastrozole will be derived, in months, as follows:

(last dose date - first dose date +1) / (365.25/12)

# 3.6 Quality of Life (QoL) questionnaires

FACT-B scores will be derived as described in section 3.4 of the main SAP

EQ-5D scores will be derived as described in section 3.5 of the main SAP.

#### 4. ANALYSIS METHODS

### 4.1 General principles

General principles of the analysis methods are unchanged from section 4.1 of the main SAP.

### 4.1.1 Multiple testing strategy

The key secondary endpoints of OS, and ORR will be tested using a multiple testing procedure (MTP) with an alpha-splitting and recycling strategy (<u>Burman et al 2009</u>). With this approach, the endpoints of OS, and ORR will be tested in a pre-defined order as shown below. The secondary endpoints of CBR, EDoR, EDoCB, FACT-B and EQ-5D will not be included in this MTP.

Figure 1 Multiple testing procedure



The primary endpoint (PFS) was tested at a single time point when 309 progression events have occurred (143 in the fulvestrant group and 232 in the anastrozole group). The secondary endpoints of OS and ORR were tested in the MTP using a weighted proportion of alpha (test mass; the total test mass equals alpha) and test mass that became available after each rejected hypothesis was recycled to secondary endpoints not yet rejected. This testing procedure stopped when the entire test mass was allocated to non-rejected endpoints. Implementation of this pre-defined ordered testing procedure included recycling, strongly controlled the Type I error at 2.5% (1-sided), amongst the primary (PFS) and the key secondary (OS and ORR) endpoints.

PFS and ORR were analysed at one time-point only. However, OS will be analysed on two occasions; at the time of the analysis of PFS and also at a later time-point when it is estimated that at least 65% of patients have died and at least 8 years have passed since the last patient was enrolled (originally planned for 50%). The available alpha will be controlled amongst the two OS analyses by using the Lan DeMets (Lan and DeMets 1983) spending function that approximates an O'Brien Fleming approach, where the significance level applied at the interim (i.e., at the time of formal PFS and ORR analysis) is dependent upon the proportion of information available. This proportion of information was calculated at the interim using the data available at that time.

Using the allocated  $\alpha$ =2% according to the MTP (ORR was not significant; one-sided p-value = 0.3645), the following was the case for the OS interim analysis:

- 142 deaths (out of the total of 462 patients recruited into the trial) occurred.
- The final OS analysis is planned for when it is estimated that at least 65% of patients have died and at least 8 years have passed since the last patient was enrolled (originally planned for 50%).
- Therefore, at the time of the interim OS analysis, it was thought that 0.6147 of the full death information (142/231 deaths) was available and the 1-sided significance level applied for the OS interim analysis was 0.00301.
- The interim OS was not statistically significant, (one-sided p-value=0.2138), therefore none of the 2% of alpha was recycled to ORR (as ORR is analysed at one time-point only).

ORR was assessed using  $\alpha$ =0.5%.

At the time of the final OS follow up analysis where at least 65% of patients have died and at least 8 years have passed since the last patient was enrolled, on the assumption that this will be conducted when 310 deaths have been observed, the one-sided significance level will be 1.845%.

#### 4.2 Analysis methods

### 4.2.1 Disposition and anti-cancer therapy

The following outputs will be produced, including all data from baseline of the main study until DCO for the follow-up analysis

| Shell<br>reference | Reference from<br>PFS analysis | Title | Notes |
|---|---|---|---|
| CCI | | Patient disposition | All patients |
| | | Important protocol deviations | Intention to treat analysis set |
| | | Disallowed concomitant<br>medication during study<br>treatment | Intention to treat analysis set |
| | | Disallowed<br>bisphosphonate/Denosumab<br>therapy during study<br>treatment | Intention to treat analysis set |
| | | All allowed concomitant<br>medications during study<br>treatment | Intention to treat analysis set |

| CCI | Post-<br>discontinuation disease-<br>related anticancer therapy | Intention to treat analysis set |
|---|---|---|
| | Discontinued subjects | All patients |
| | Subjects ongoing study at data cut-off | Intention to treat analysis set |
| | Subjects with important protocol deviations | Intention to treat analysis set |
| | Medication on entry and during the study | Intention to treat analysis set |

#### 4.2.2 Overall survival

The following OS tables, listings and figures (TLFs) will be produced, with amendments as noted below. All OS outputs will include the footnote:

Patients not known to have died are censored at the date they were last known to be alive, as recorded on the survival status CRF.

| Shell<br>reference | Reference from<br>PFS analysis | Title | Notes |
|---|---|---|---|
| CCI | | Survival status at the time<br>of the OS analysis,<br>secondary analysis at 65%<br>OS maturity <sup>1</sup> | |
| | | Median overall survival at<br>the time of the OS<br>analysis, secondary<br>analysis at 65% OS | Quartiles (if reached) and<br>median (50 <sup>th</sup> percentile)<br>OS will be summarised |
| | | maturity <sup>1</sup> | Percentage OS at 6<br>monthly intervals up to<br>an appropriate time point<br>will be summarised |
| | | Overall survival, Stratified<br>log-rank test, secondary<br>analysis at 65% OS<br>maturity <sup>1</sup> | |

Sensitivity analysis of overall survival, Cox proportional hazards regression model, secondary analysis at 65% OS maturity<sup>1</sup> Overall survival, Stratified Subgroups are defined in log-rank test, subgroup section 4.2.1.2 of the analysis, secondary main SAP analysis at 65% OS maturity<sup>1</sup> Overall survival, Stratified Geographical region log-rank test, geographical subgroups are defined in section 4.2.1.2 of the region subgroup analysis, secondary analysis at 65% main SAP OS maturity<sup>1</sup> Summary of total follow-Follow-up is defined as up (months) for OS of all the duration of follow-up patients, secondary is defined as the number analysis at 65% OS of months from maturity<sup>1</sup> randomisation to death or last contact Patients censored for OS A patient unknown to be at more than 12 weeks alive or dead at the time before secondary analysis of the DCO will be at 65% OS maturity<sup>1</sup> censored at the time they were last known to be alive (this differs to the programming notes in the shell) Overall survival at the time of secondary analysis at 65% OS maturity<sup>1</sup>, Kaplan-Meier plot Subgroups are defined in Overall survival at the section 4.2.1.2 of the time of secondary analysis main SAP at 65% OS maturity<sup>1</sup>,

Kaplan-Meier plot (for

subgroup: xxx)

| CCI | Overall survival at the time of secondary analysis after 65% of patients have died <sup>1</sup> , Kaplan-Meier plot (for subgroup: Geographic region: xxx) | Geographical region<br>subgroups are defined in<br>section 4.2.1.2 of the<br>main SAP |
|---|---|---|
| | Time to censoring for<br>secondary analysis after<br>65% of patients have<br>died <sup>1</sup> , Kaplan Meier plot | |
| | Overall survival at the<br>time of secondary analysis<br>after 65% of patients have<br>died <sup>1</sup> , Forest plot, by<br>subgroup | |
| | Overall survival at the time of secondary analysis after 65% of patients have died <sup>1</sup> , Forest plot, by geographical region subgroup | |
| | Overall survival status at<br>time of secondary analysis<br>at 65% OS maturity <sup>1</sup> | |

At least 65% of patients have died and at least 8 years have passed since the last patient was enrolled

# 4.2.3 Best response to first subsequent breast cancer therapy

Best overall response subsequent to the first subsequent cancer therapy will be summarised as follows:

| Shell<br>reference | Reference from PFS analysis | Title | Notes |
|---|---|---|---|
| NA | NA | Summary of best overall<br>tumour response to the first<br>subsequent therapy | CCI |

| NA | NA | Summary of best overall tumour response to the first subsequent therapy by subsequent therapy |
|---|---|---|
| CCI | | Listing of systemic<br>anticancer therapy post<br>randomisation |





# 4.2.4 Exposure to study drug

Total and actual treatment durations will be summarised by treatment group, from the baseline of the main study until DCO for the follow-up analysis.

| Shell<br>reference | Reference from PFS analysis | Title |
|---|---|---|
| CCI | | Duration of exposure |
| | | Study drug administration - fulvestrant and anastrozole |
| | | Duration of exposure |

## 4.2.5 Safety

Deaths and SAEs, from baseline of the main study until DCO for the follow-up analysis, will be listed for each patient and summarised by treatment received according to the system organ class (SOC) and preferred term (PT).

| Shell<br>reference | Reference from<br>PFS analysis | Title |
|--------------------|--------------------------------|------------|
| CCI | | All Deaths |

| CCI | Serious Adverse Events with outcome of death by system organ class and preferred term |
|---|---|
| | Serious Adverse Events with outcome of death, causally related to study treatment |
| | Listing of deaths |
| | Serious Adverse Events with outcome of death - key patient information |
| | Serious adverse events, by system organ class and preferred term |
| | Serious adverse events, causing discontinuation from treatment, by system organ class and preferred term |
| | Serious adverse events, causally related to study<br>treatment by system organ class and preferred term |
| | Serious adverse events, leading to study treatment discontinuation, causally related to study treatment |
| | Serious adverse events - Listing of key information for SAEs |
| | Listing of serious adverse events (1) |
| | Listing of serious adverse events (2) |
| | Listing of serious adverse events (3) |

## 4.2.6 Quality of Life (QoL) questionnaires

### 4.2.6.1 FACT-B

All visits from the baseline of the main study until DCO for the follow-up analysis will be included in the summary of the FACT-B scores; specifically Trial Outcome Index (TOI), total FACT-B. Individual subscale scores will not be summarised in the follow-up analysis. The analysis of time to deterioration of TOI and FACT-B total score will be as outlined for the main SAP.

| Shell<br>reference | Reference from PFS analysis | Title | Notes |
|---|---|---|---|
| CCI | | Compliance with FACT-B by time point. | CCI |
| - | | FACT-B total score over time | |

| | _ | |
|-----|--------------------------------------------|---------------|
| CCI | Trial outcome index (TOI) score over | |
| | time | |
| | FACT-B total score - change from | |
| | baseline and categories of change from | |
| | baseline | |
| | Trial outcome index (TOI) score over | |
| | time - change from baseline and | |
| | categories of change from baseline | |
| | o o | |
| | FACT-B total score and TOI score time | |
| | to deterioration (months) | |
| | , , | |
| | Analysis of time to deterioration of | Remove the p- |
| | FACT-B total score | value |
| | Analysis of time to deterioration of trial | Remove the p- |
| | outcome index score | value |
| | Mean (+/- SD) FACT-B total score | |
| | across timepoints, by treatment group | |
| _ | | |
| | Mean (+/- SD) trial outcome index (TOI) | |
| | score across timepoints, by treatment | |
| | group | |
| _ | | |
| | Mean (+/- SD) FACT-B total score | |
| | change from baseline across timepoints, | |
| | by treatment group | |
| | Mean (+/- SD) trial outcome index (TOI) | |
| | change from baseline across timepoints, | |
| | by treatment group | |
| _ | | |
| | Kaplan-Meier plot for time to | |
| | deterioration (months) - FACT-B total | |
| | score | |
| | Kaplan-Meier plot for time to | |
| | deterioration (months) of TOI | |
| - | | |
| | Review of patient reported outcomes | |
| | questionnaire - FACT-B | |
| - | 7.7. | |
| | Listing of total score by FACT-B | |
| | domain | |

### 4.2.6.2 EQ-5D

All visits from the baseline of the main study until DCO for the follow-up analysis will be included in the summary of EQ-5D individual questions and combined health score with be listed. VAS score and UK health state utility values and change from baseline will be listed and summarised. VAS score and health state combined score compliance rates will also be summarised similarly to FACT-B.

| Shell<br>reference | Reference from<br>PFS analysis | Title |
|---|---|---|
| CCI | | EQ-5D questionnaire - (VAS) score and health state combined score compliance rate by time point |
| | | EQ-5D questionnaire - (VAS) score and UK health state utility value - summary scores |
| | | EQ-5D questionnaire - (VAS) score and UK health state utility value - change from baseline |
| | | Review of patient reported outcomes questionnaire - EQ-5D |
| | | Listing of EQ-5D questionnaire - individual questions and health state combined score |
| | | Listing of EQ-5D questionnaire - health scores |
| | | Listing of EQ-5D questionnaire - health scores change from baseline |

#### 5. REFERENCES

#### Burman et al 2009

Burman CF, Sonesson C, Guilbaud O. A recycling framework for the construction of Bonferroni-based multiple tests. Statistics in Medicine 2009:28;739–761.

#### Lan and DeMets 1983

Lan KKG, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika 1983;70;3:659-63.

# SIGNATURE PAGE

This is a representation of an electronic record that was signed electronically and this page is the manifestation of the electronic signature

| Document Name: d699bc00001-sap-addendum-edition-2 | | |
|---|---|---|
| Document Title: | Statistical Analysis Plan Addendum Edition 2 | |
| Document ID: | CCI | |
| Version Label: | 2.0 CURRENT LATEST APPROVED | |
| Server Date<br>(dd-MMM-yyyy HH:mm 'UTC'Z) | Signed by | Meaning of Signature |
| 11-May-2022 17:05 UTC | PPD | Author Approval |

Notes: (1) CCI